CLINICAL TRIAL: NCT03821571
Title: Evaluation of Cerebral Small Vessel Disease in Patient With Primary Aldosteronism
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201811039RIND
Record Dates: First submitted 2019-01-24; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Evaluation of Cerebral Small Vessel Disease in Patient With Primary Aldosteronism
Keywords: Hypertension,primary aldosteronism
MeSH Terms: conditions — Hypertension; Hyperaldosteronism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with primary aldosteronism (Experimental): Brain MRI with T1WI, T2WI, FLAIR, thin-sliced T1WI, DWI, TOF, and blood sensitive sequence (SWI) will be performed.
  Interventions: Diagnostic Test: Brain MRI
- Patient with essential hypertension (Active Comparator): Brain MRI with T1WI, T2WI, FLAIR, thin-sliced T1WI, DWI, TOF, and blood sensitive sequence (SWI) will be performed.
  Interventions: Diagnostic Test: Brain MRI

INTERVENTIONS:
Diagnostic Test: Brain MRI — Brain MRI with blood sensitive sequence (SWI) will be performed to all enrolled patients.

SUMMARY:
Hypertension is known to be the major risk factor for stroke. The most common cause of secondary hypertension, primary aldosteronism (PA), is characterized by the excessive secretion of aldosterone and is related to hypertension and hypokalemia. PA accounts for 3-10 % of hypertensive patients, and a higher incidence of vascular complications compared to patients with essential hypertension was observed in several studies. The vascular injury from excessive aldosterone can occur via oxidative stress and collagen remodeling, causing endothelial dysfunction and fibrosis in the vasculature.

The association between cerebral small vessel disease (cSVD) and hypertension has been well studies in the past decades. However, not much study has focused on the cSVD burden in patient with PA. The goal of this study is to understand the features of cSVD in patients with PA and for the purpose of understanding the underlying pathophysiology of cerebrovascular injury in this particular patient group.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-90 years-old
* patient with primary aldosteronism or healthy control
* consciousness clear
* willing to receive brain MRI

Exclusion Criteria:

* renal failure or Creatinine > 2mg/dl
* coagulopathy or hepatic insufficiency
* unstable vital sign under inotropic agents
* pregnancy
* metal implant or cardiac pacemaker
* major brain surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-25 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebrovascular reactivity | During the brain MRI
  Cerebrovascular reactivity measured by MRI under primary aldosteronism

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Hsi Tsai, MD, Principal Investigator — Bei-Hu branch, National Taiwan University Hospital
Locations (1):
- Bei-Hu Branch, National Taiwan University Hospital, Taipei, Taiwan